CLINICAL TRIAL: NCT04009564
Title: Investigating the Acute Effects of Mood and Cognitive Performance Following the Administration of a Coffee Made of Date Seeds on Healthy Young Volunteers.
Brief Title: Effect of Date Seeds Coffee on Mood and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DSCPM
Record Dates: First submitted 2018-12-19; First posted 2019-07-05 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2019-07

CONDITIONS: Health Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Date seeds filtered coffee (Experimental): Each participant will consume this arm in a visit has been allocated by Latin Square randomisation order: 45 g of date seeds coffee in 280 ml of boiled water, coffee flavour and brown food colouring ( made using a filter coffee machine). it will be served in a paper cup with lid
  Interventions: Dietary Supplement: Date coffee
- Normal filtered coffee (Experimental): Each participant will consume this arm in a visit has been allocated by Latin Square randomisation order: 6 g of coffee in 280 ml of boiled water (made using a filter coffee machine) it will be served in a paper cup with lid
  Interventions: Dietary Supplement: Normal coffee
- Placebo (Placebo Comparator): Each participant will consume this arm in a visit has been allocated by Latin Square randomisation order: 280 of boiled water, coffee flavour and brown food colouring it will be served in a paper cup with lid
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Date coffee — 45 g of date seeds coffee in 280 ml of water
  Arms: Date seeds filtered coffee
Dietary Supplement: Normal coffee — 6 g of normal coffee in 280ml of water
  Arms: Normal filtered coffee
Dietary Supplement: Placebo — water, food colouring and coffee flavouring
  Arms: Placebo

SUMMARY:
Limited utilizations of date seeds have previously been explored, and so previously wastage has often been the normality. However, research now indicates that several fruit seeds contain higher concentrations of beneficial total phytochemicals within their seeds in comparison to the flesh. As well as high nutritional values of date seeds for fibre, protein and micronutrients, this increased phytochemical content has been proven to be true for date seeds, with mainly phenolic acids (24.6 g k GAE) 3 and total flavonoids (3.67 g k RE). With the seeds presently being used to produce new coffee products, it raises questions on whether consumption of date seeds can alter mood and cognitive behaviour and therefore research into investigate the acute effect of date seeds coffee on mood and cognitive function on healthy young volunteers. However, to the best of the research team knowledge, this is the first human trial to investigate these effects.

DETAILED DESCRIPTION:
Introduction

Seeds of the date palm (P. dactylifera) are a very rich source of bioactive compounds, thus constituting strong candidates for functional food additives and nutraceuticals. Many promising results were observed when the effect of date flesh and seeds consumption have been studied in animals, for their role as either a protective1 against neurodegenerative 2,4,5 diseases, or as a cure for it 2. Most of the observed effects were attributed to the antioxidant and anti-inflammatory properties in dates flesh and seeds fruit due to it high content of phenolic compounds 3.

Rational For years, date seeds were considered a waste, having no other uses except for feeding animals. However, as has already been demonstrated in other fruits and corresponding seeds, total phytochemical content of the date seeds was higher than in the edible flesh9. Date seeds have also been shown to have an excellent nutritional quality due to high amounts of fibre (676-742 g/kg) 3 depending on variety, considerable amounts of minerals, vitamins, lipids and protein. Additionally, date seeds were shown to be rich in antioxidants containing mainly phenolic acids (24.6 g k Gallic Acid equivalent) 3 and total flavonoids (3.67 g k Rutin Equivalent).

Nowadays, and on sight of the aforementioned findings, date seeds are used to make a new coffee product. This ''coffee alternative'' is commercially available and is becoming more popular.

Although, many studies have demonstrated that date seeds possess high antioxidant activities, due to their high content of flavonoids and phenolic compounds, no human trial has investigated the effect of the consumption of date seeds on humans and especially on mood and cognitive behaviour. Therefore, this study, for the first time, to the best of the research team knowledge will investigate the acute effect of date seeds coffee on mood and cognitive function on healthy young volunteers.

Aim The aim of this study is to investigate the acute effects of a coffee made of date seeds on mood and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

Healthy young volunteers age between 18 to 35

Exclusion Criteria:

Participants will be ineligible to participate in the study if any of the following apply:

1. Have a BMI above 35kg/m2
2. Smokers or tobacco product consumers which includes electronic cigarettes
3. Are taking any illicit or prescribed drugs.
4. Have a history of, or currently, abuse alcohol
5. Have a history of dyslexia, ADHD, learning difficulties or colour blindness,
6. Females who are pregnant, lactating or seeking to become pregnant, or are at risk of pregnancy as they to do not use birth control measures
7. Have allergies to any food product.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The average of the change in 9 cognitive indexes including: Attentional Intensity, Sustained Attention, Attentional Fluctuation, Memory Retrieval Speed, Cognitive Reaction Time, Working Memory Capacity, Episodic Memory Capacity, Quality of Memory | Change from baseline at 45 minutes post dose and at 90 minutes post dose for each visit
  Cog-track an online set of nine cognitive tests (www.wesnes.com).

SECONDARY OUTCOMES:
Change in Caffeine consumption using caffeine consumption questionnaire | Change form Baseline for each visit only
  A paper based questionnaire developed by Erika Bühler et al., 2014. At the screening visit and on each study day participants will be asked to complete the table in order to build a picture of their individual caffeine habits
Caffeine research Visual Analogue Scales | Change from baseline 45 minutes post dose and at 90 minutes post dose.
  A caffeine research Visual Analogue Scales which comprises of 7 scales (relaxed, alert, jittery, tired, tense, headache and overall mood).
Change in Mood using Bond Lader Visual Analogue Scales | Change from baseline 45 minutes post dose and at 90 minutes post dose.
  This widely used set of 16 100 mm VASs yields three extensively validated factor scores: alertness, calmness and contentment.

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided